CLINICAL TRIAL: NCT03500484
Title: Effect of Liraglutide on Neural Responses to High Fructose Corn Syrup in Individuals With Obesity.
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The study was initially paused due to COVID restrictions and then when able to resume, there was no longer funding.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2000022407
Record Dates: First submitted 2018-04-09; First posted 2018-04-18 (Actual); Results first posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Obesity, Childhood; Neural Development
MeSH Terms: conditions — Pediatric Obesity | interventions — Liraglutide; Glucagon-Like Peptide 1

STUDY DESIGN:
Intervention Model Description: 15 control and 30 obese subjects
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- obese subjects (Experimental): Subjects will self-administer Liraglutide once daily for 12 weeks.
  Interventions: Drug: Liraglutide
- lean subjects (No Intervention): no intervention

INTERVENTIONS:
Drug: Liraglutide — Liraglutide will be supplied in the following package sizes containing disposable, pre-filled, multidose pens. Each individual pen delivers doses of 0.6 mg, 1.2 mg, 1.8 mg, 2.4 mg or 3 mg (6 mg/mL, 3 mL). Liraglutide will be self-administered daily for 12 weeks under the following regimen: 0.6mg for 1 week, 1.2mg for 1 week, 1.8mg for 1 week, 2.4mg for 1 week, 3.0mg until week 12.
  Other Names: Glucagon-like peptide 1
  Arms: obese subjects

SUMMARY:
To study the effects of liraglutide on neural responses to high fructose corn syrup (HFCS) in individuals with obesity.

DETAILED DESCRIPTION:
Adolescents are the highest consumers of sugar sweetened beverages (SSB) potentially because their developing brains are most susceptible to the rewarding neural effects of sugar consumption. Thus, we specifically target this population (adolescents) to understand neural mechanisms involved in excess sugar consumption which predisposes to the development of obesity, prediabetes, and type 2 diabetes.

Upon results entry, the data elements in protocol section of this record were updated to reflect the appropriate study phase and primary purpose that was inadvertently mischaracterized at the time of registration. One of the secondary outcomes was removed because it was a duplicate of the second primary outcome.

ELIGIBILITY:
Inclusion Criteria:

1. 18-39 years old
2. Lean (BMI 18.5-24.9 kg/m2) with normoglycemia
3. Obese (BMI 30-45 kg/m2) with or without prediabetes
4. Weight stable
5. Right handed
6. Able to read and write in English
7. Able to provide written and verbal informed consent

Exclusion Criteria:

1. Current active participation in a weight loss program or weight loss of >=10% of total body weight during the previous 6 months
2. Prior bariatric surgery or current gastric balloon
3. Weight >440lbs or waist circumference >142cm
4. Following a vegetarian/vegan diet or dieting/restricting food
5. Significant medical condition
6. Current use of weight-loss medications or supplements, psychiatric medications or anti- hyperglycemic medications
7. History of or family history of multiple endocrine neoplasia type 1 (MEN-I) or medullary thyroid cancer, alcoholism, or previous history of pancreatitis
8. Females who are pregnant or lactating, or who are unwilling to use proper contraception or remain abstinent,
9. Claustrophobia that would interfere with MRI or metal in their body that would pose a risk in the MRI.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ania Jastreboff, Phd,MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Obesity: Subjects self-administer Liraglutide once daily for 12 weeks.
  Liraglutide: Liraglutide supplied in the following package sizes containing disposable, pre-filled, multidose pens. Each individual pen delivers doses of 0.6 mg, 1.2 mg, 1.8 mg, 2.4 mg or 3 mg (6 mg/mL, 3 mL). Liraglutide self-administered daily for 12 weeks under the following regimen: 0.6mg for 1 week, 1.2mg for 1 week, 1.8mg for 1 week, 2.4mg for 1 week, 3.0mg until week 12.
- Participants Who Are Lean: no intervention
Period: Overall Study
Arm/Group | Participants With Obesity | Participants Who Are Lean
Started | 8 | 5
Completed | 4 | 5
Not Completed | 4 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Could not be scanned or followed up due to COVID | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Obese Subjects | Lean Subjects | Total
Number analyzed (Participants) | 8 | 5 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (5.5) | 21.2 (1.9) | 24.2 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 1 | 3
  African American | 3 | 1 | 4
  Hispanic | 3 | 0 | 3
  Asian | 0 | 2 | 2
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 5 | 13
Years of Education [Mean (Standard Deviation); unit: years] | 14 (2.9) | 15 (1.8) | 14 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Brain Response in Obese Young Adults Who Drink Sugar Sweetened Beverages.
Description: To investigate brain response (using fMRI) to acute consumption of sugar sweetened beverages in obese prediabetic adolescents/young adults (age 18-39 yrs), increase in cerebral blood flow was monitored in participants as a binary outcome (increase/no increase).
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Groups:
- Participants With Obesity: Subjects self-administer Liraglutide once daily for 12 weeks.
  Liraglutide: Liraglutide supplied in the following package sizes containing disposable, pre-filled, multidose pens. Each individual pen delivers doses of 0.6 mg, 1.2 mg, 1.8 mg, 2.4 mg or 3 mg (6 mg/mL, 3 mL). Liraglutide will be self-administered daily for 12 weeks under the following regimen: 0.6mg for 1 week, 1.2mg for 1 week, 1.8mg for 1 week, 2.4mg for 1 week, 3.0mg until week 12.
Arm/Group | Participants With Obesity | Participants Who Are Lean
Number analyzed (Participants) | 8 | 5
Participants
  Increase in cerebral blood flow in the caudate, putamen and insula | 8 | 0
  No increase in cerebral blood flow in the caudate, putamen and insula | 0 | 5

2. Primary Outcome: Change in Brain Response in Obese Young Adults Who Drink Sugar Sweetened Beverages.
Description: To investigate brain response (using fMRI) to acute consumption of sugar sweetened drinks in obese prediabetic adolescents/young adults (age 18-39 yrs). Measurement at 1 week was compared to measurement at 12 weeks. Increased blood flow in thalamus was monitored in participants as a binary outcome (increase/no increase).
Time Frame: 1 week and 12 weeks
Population: 12 week follow up only took place in participants with obesity in matched cases.
Measure: Count of Participants; unit: Participants
Groups:
- Participants With Obesity: Subjects will self-administer Liraglutide once daily for 12 weeks.
  Liraglutide: Liraglutide will be supplied in the following package sizes containing disposable, pre-filled, multidose pens. Each individual pen delivers doses of 0.6 mg, 1.2 mg, 1.8 mg, 2.4 mg or 3 mg (6 mg/mL, 3 mL). Liraglutide will be self-administered daily for 12 weeks under the following regimen: 0.6mg for 1 week, 1.2mg for 1 week, 1.8mg for 1 week, 2.4mg for 1 week, 3.0mg until week 12.
Arm/Group | Participants With Obesity
Number analyzed (Participants) | 4
Participants
  Increased blood flow in thalamus at 1 week | 0
  Increased blood flow in thalamus at 12 weeks | 4

3. Other Pre Specified Outcome: To Investigate the Role of Specific Metabolic/Hormonal Responses in the Setting of Liraglutide Treatment, in Affecting Neural Responses to Sugar Ingestion.
Description: To investigate the role of specific metabolic/hormonal responses in the setting of liraglutide treatment, in affecting neural responses to sugar ingestion. Metabolic response is represented by the whole-body insulin sensitivity index (WBISI). The Oral Glucose Tolerance Test (OGTT) were performed at Baseline and Week 12. Insulin Sensitivity was measured by obtaining glucose and insulin levels in a fasting state and at 2 hours after administration of oral glucose load. Matsuda index = 10,000/SQRT [glucose concentration (mg/dL) (fasting)*insulin concentration (uIU/mL) (fasting)*glucose concentration (mg/dL) (2 hours after glucose load)*insulin concentration (uIU/mL) (2 hours after glucose load)], with higher numbers indicating better insulin sensitivity.
Time Frame: 1 week and 12 weeks
Population: 12 week follow up only took place in participants with obesity in matched cases.
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Participants With Obesity
Number analyzed (Participants) | 4
Index
  1 Week | 3.54 (2.05)
  12 Weeks | 4.08 (3.58)

ADVERSE EVENTS:
Time Frame: 12-16 weeks
Description: definition used do not differ from clinicaltrials.gov
Groups:
- Participants With Obesity: Subjects self-administer Liraglutide once daily for 12 weeks.
  Liraglutide: Liraglutide be supplied in the following package sizes containing disposable, pre-filled, multidose pens. Each individual pen delivers doses of 0.6 mg, 1.2 mg, 1.8 mg, 2.4 mg or 3 mg (6 mg/mL, 3 mL). Liraglutide will be self-administered daily for 12 weeks under the following regimen: 0.6mg for 1 week, 1.2mg for 1 week, 1.8mg for 1 week, 2.4mg for 1 week, 3.0mg until week 12.
Arm/Group | Participants With Obesity | Participants Who Are Lean
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/5
Other Adverse Events (participants affected / at risk) | 3/8 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Obesity (N=8) | Participants Who Are Lean (N=5)
gastrointestinal side effects and patient dx with sarcoidosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
rash near injection area (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT03500484/Prot_SAP_000.pdf